CLINICAL TRIAL: NCT03773237
Title: Randomized Prospective Trial Comparing Intralipid Versus SMOFlipid in New HPN Patients.
Brief Title: Intralipid Versus SMOFlipid in HPN Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17-001403
Record Dates: First submitted 2018-11-12; First posted 2018-12-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-10

CONDITIONS: Short Bowel Syndrome; Intestinal Fistula; Crohn Disease; Intestinal Obstruction
Keywords: SMOF; Intralipid; Mixed oil emulsion; Intestinal failure; HPN
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Fistula; Crohn Disease; Intestinal Obstruction; Intestinal Failure | interventions — SMOFlipid; soybean oil, phospholipid emulsion

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization list will be generated using http://www.randomization.com and blinded at enrollment using supplement codes. The study coordinator will hold the randomization codes and will be revealed to the investigators only after the statistical analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMOFLipid (Active Comparator): SMOFlipid is a lipid emulsion that contains a combination of soybean oil, medium chain triglycerides, olive oil, and fish oil.
  Interventions: Dietary Supplement: SMOFLipid
- IntraLipid (Active Comparator): Intralipid is a lipid emulsion that contains soybean oil
  Interventions: Dietary Supplement: Intralipid

INTERVENTIONS:
Dietary Supplement: SMOFLipid — SMOFLipid will be given to HPN patients to assess the benefits or adverse effects compared to Intralipid.
  Arms: SMOFLipid
Dietary Supplement: Intralipid — Intralipid will be given to HPN patients to assess the benefits or adverse effects compared to SMOFlipid
  Arms: IntraLipid

SUMMARY:
This study will randomize all patients who are new to the Mayo Clinic HPN team to either standard lipid emulsion (Intralipid) or SMOFLipid.

DETAILED DESCRIPTION:
Primary aim is to assess the impact to direct/indirect bilirubin.

Secondary aims will be to assess impact to other liver function studies, metabolic parameters, inflammatory marker, body weight, ability to meet caloric needs through TPN, and ability to obtain appropriate macronutrient composition.

ELIGIBILITY:
Inclusion Criteria:

* Newly initiated Mayo Clinic HPN patient
* Able to provide informed consent
* Anticipated duration of HPN greater than 3 months,
* Infusion company is able to provide Smoflipid

Exclusion Criteria:

* Age less than 18 years
* Pregnant and lactating women
* Failure to provide consent
* Patients with underlying liver dysfunction (defined as liver function studies equal to or more than 2 times upper limit of normal) or pathology as determined by primary investigator
* Patients with active malignancy
* Patients who are deemed to be on HPN for less than three months
* Patients who have previous proven addiction and dependence to alcohol/ heavy alcohol AND consumption/active use reported during last 12 months.
* Known hypersensitivity to fish, egg, soybean, or peanut protein, or to any of the active ingredients or excipients in Smoflipid
* Patients who will not be managed by the Mayo Clinic HPN team
* Patients who have active infection (as determined by the clinician) at the time of enrollment.
* Patients who have received Smoflipid greater than 4 weeks in the last 12 months prior to enrollment.
* Patients who have been on TPN greater than 4 weeks in the last 12 months prior to enrollment.
* Enrolled in another interventional study.
* Severe hyperlipidemia or severe disorders of lipid metabolism with serum triglycerides more than 1,000 mg/dL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Direct/Indirect Bilirubin Change is assessed | At 12 weeks weeks
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet S Mundi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials